CLINICAL TRIAL: NCT03060954
Title: A Multicentre, Controlled, Randomised, Single-blind, Two-armed Trial Evaluating the Visual Performance, Quality of Vision and Subjective Outcomes After Bilateral Implantation of MINI WELL Ready® or FineVision® in Patients With Cataract Surgery.
Brief Title: Non-Inferiority Study Comparing MINI WELL READY® and FineVision® in Patients With Cataract Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical study is closed to further enrolment based on the lack of perceived need to compare the study device with the control device.
Sponsor: SIFI SpA (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PSM29
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINI WELL READY ® (Experimental): BILATERAL IMPLANTATION OF MINI WELL READY®, A PROGRESSIVE EXTENDED DEPTH OF FOCUS INTRAOCULAR LENS IN PATIENTS WITH CATARACT SURGERY
  Interventions: Device: MINI WELL READY ®
- FineVision ® (Other): FINE VISION®, A TRIFOCAL INTRAOCULAR LENS IMPLANTATION IN PATIENTS WITH CATARACT SURGERY
  Interventions: Device: FINE VISION®

INTERVENTIONS:
Device: MINI WELL READY ® — BILATERAL IMPLANTATION OF MINI WELL READY®, A PROGRESSIVE EXTENDED DEPTH OF FOCUS INTRAOCULAR LENS IN PATIENTS WITH CATARACT SURGERY
  Arms: MINI WELL READY ®
Device: FINE VISION® — FINE VISION®, A TRIFOCAL INTRAOCULAR LENS IMPLANTATION IN PATIENTS WITH CATARACT SURGERY
  Arms: FineVision ®

SUMMARY:
Interventional, Multicentre, controlled, randomized, single blind, twoarmed non-inferiority trial

DETAILED DESCRIPTION:
To evaluate the non-inferiority of the progressive extended depth of focus Intraocular Lens MINI WELL READY® in terms of visual performance, quality of vision and subjective outcomes versus the trifocal Intraocular Lens FineVision® after a follow up period of 2-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bilateral cataract surgery required, no other ocular comorbidities
* Healthy corneas, not treated surgically
* Available for second-eye surgery within 1 week of the initial operation
* Spherical refraction between -8.00D and +6.00D
* Willing to adhere to the study visit schedule
* Normal anterior and posterior segments
* Clear intraocular media - other than cataract
* To benefit from a social security system before being enrolled
* Written informed consent consistent with local regulation research in human subjects

Exclusion Criteria:

* Any previous history of ocular trauma or prior ocular surgery (including previous cataract surgery and CLRIs)
* Ocular comorbidities determining potential postoperative Visual Acuity less than 0.50 decimal (0.3 logMAR)
* Expected to require retinal laser treatment
* A history of retinal detachment or predisposition for such disorder
* Psudoexfoliation
* Abnormal pupil size and position
* Pupil size > 7 mm under mesopic condition
* Use of contact lenses 30 days before the preoperative visit
* Corneal warpage (e.g. Keratoconus, Pellucid Marginal Corneal Degeneration or Keratoglobus)
* Corneal astigmatism greater than 0.75D
* Zonular laxicity
* Absence of adequate capsular support for the implant of the intraocular lens in the capsular bag
* Microphthalmus
* Active ocular disease in the operative eye, for example, chronic uveitis, proliferative diabetic retinopathy, chronic glaucoma unresponsive to medication, corneal decompensation and corneal endothelial cell insufficiency (such as Fuch's endothelial dystrophy)
* Suspected microbial infection
* Irregularities and capsulorexis decentralization
* Surgical difficulties that may increase the risk of complications such as persistent bleeding, significant iris damage, an uncontrollable intraocular hypertonia, or damage due to significant vitreous loss
* Patients in whom the intraocular lens may interfere with the ability to observe, diagnose or treat diseases of the posterior segment
* Patients in whom neither the posterior capsule nor the zonula can provide adequate support to the lens
* Subjects with any systemic disease that could increase operative risk or confound the outcome
* Pregnant or lactating or planning a pregnancy at the time of enrolment
* Vulnerable subjects (children <18 years, people in guardianship or trusteeship or inability to give an informed consent)
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Defocus curve - binocular | 6 months
  Defocus curve assessment

OTHER OUTCOMES:
Refraction | 6 months
  Ocular refraction evaluation
Visual Acuity Evaluation | 6 months
  Uncorrected Distance Visual Acuity (UDVA)
Visual Acuity Evaluation | 6 months
  Corrected Distance Visual Acuity (CDVA) Uncorrected Intermediate Visual Acuity (UIVA)
Visual Acuity Evaluation | 6 months
  Distance Corrected Intermediate Visual Acuity (DCIVA)
Visual Acuity Evaluation | 6 months
  Uncorrected Near Visual Acuity (UNVA)
Visual Acuity Evaluation | 6 months
  Distance Corrected Near Visual Acuity (DCNVA)
Reading speed | 6 months
  Reading speed performance
Halometry | 6 months
  Halos evaluation
Contrast sensitivity | 6 months
  Contrast sensitivity evaluation
Subject satisfaction questionnaire - VF-11R | 6 months
  Subject satisfaction questionnaire - VF-11R "revised version":
  Annex A: Subject's glasses independence and light dependence Annex B: Quality of Vision (QoV) questionnaire
Operative Complications / Postoperative Complications / Adverse Event Assessment | 6 months
  Assessment of Operative Complications, Postoperative Complications, Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Stivale, Study Director — SIFI SpA
Locations (2):
- France (2):
  - Ophtalmologie Hôpital Morvan, Brest
  - Clinique Juge, Marseille

IPD SHARING:
Plan to Share IPD: Yes